CLINICAL TRIAL: NCT00788658
Title: Cognitive Behavior Therapy (CBT) as Compared With Standard Therapy for Patients With IBS and Other Functional Gastrointestinal Disorders
Brief Title: Cognitive Behaviour Therapy for Patients With IBS
Acronym: EFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ram Dickman, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC 5139
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Irritable Bowel Syndrome; Constipation; Abdominal Pain; Depression
Keywords: Obstructed constipation; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Abdominal Pain; Depression | interventions — Diet Therapy; Diet; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet modifications (Placebo Comparator): Diet consultation and life style modifications for 6 sessions
  Interventions: Behavioral: Diet modifications
- Cognitive therapy (Active Comparator): 6 sessions of cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Diet modifications — Diet consultation
  Other Names: Diet
  Arms: Diet modifications
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy
  Other Names: CBT
  Arms: Cognitive therapy

SUMMARY:
Irritable bowel syndrome (IBS) affects approximately 10-15% of the adult population. This condition is characterized by abdominal pain, altered bowel habit, abdominal bloating and reduced quality of life. Options for treating IBS include pharmacotherapy, psychotherapy, hypnotherapy and cognitive behavior therapy (CBT). Available data on the effectiveness of CBT in IBS patients in Israel are scarce.

The aim of the present study is to assess effectiveness of CBT as compared with standard therapy for IBS patients in Israel The course of CBT consisted of up to six 40 min sessions, and included education about IBS and techniques to reduce focusing on symptoms and to manage stress.Standard therapy includs life style modifications.

The primary outcome measure was the score on a symptom-severity scale specific to IBS.

DETAILED DESCRIPTION:
Symptomatic treatment of patients would not be modified

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* IBS

Exclusion Criteria:

* Malignancy
* Known psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Symptom score | 3 months

SECONDARY OUTCOMES:
Quality of life assessment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ram Dickman, MD, Principal Investigator — RMC